CLINICAL TRIAL: NCT04237285
Title: Effectiveness of Inhalation Aromatherapy In Children With Burns: A Randomized Controlled Trial
Brief Title: Effectiveness of Inhalation Aromatherapy In Children With Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, ESRA ARDAHAN AKGUL, Research Assistant, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/201
Record Dates: First submitted 2020-01-14; First posted 2020-01-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Burns
Keywords: pediatric; aromatherapy
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lavender 15 (Experimental): Participant who inhalates lavender oil for 15 minutes.
  Interventions: Other: Inhalation aromatherapy
- Lavender 60 (Experimental): Participant who inhalates lavender oil for 60 minutes.
  Interventions: Other: Inhalation aromatherapy
- Jojoba (Placebo Comparator): Participant who inhalates jojoba oil for 15 minutes.
  Interventions: Other: Inhalation aromatherapy

INTERVENTIONS:
Other: Inhalation aromatherapy — Besides routine care, the Control Group was treated with jojoba oil (Simmondsia Chinensis- produced by Arifoğlu, obtained from jojoba fruits by cold squeezing method) inhalation aromatherapy 15 minutes before Hydrotherapy. Jojoba oil was used as a placebo because it had no specific odor. Besides routine care Intervention-15 Group received lavender oil (Lavandula angustifolia Miller Oleum-produced by Arifoğlu, obtained from lavender flowers by water vapor distillation method) inhalation aromatherapy 15 minutes before Hydrotherapy and besides routine care Intervention-60 Group received lavender oil inhalation aromatherapy 60 minutes before Hydrotherapy.

SUMMARY:
The study was carried out in the Pediatric Burn Unit, aged between 2 months and 7 years, with no chronic pain, second degree superficial scald burns, hydrotherapy application, no burn surgery, no pathogen growth in the burn site, the burn had not undergone epithelialization. Children receiving routine analgesic therapy were included.

Lavender oil 15 minutes, Lavender oil 60 minutes and Jojoba oil 15 minutes (Placebo group) were studied with a total of 108 children in three groups.

The children included in the study were randomized. One of the researchers measured the pain and vital signs of children before the application. 0.5 cc of aromatherapy oil, which was dripped into the gauze 15 or 60 minutes before the start of hydrotherapy and dressing, was placed 20 cm away from the child's nose. The child who inhaled the smell was hydrotherapy and dressing and then taken to bed. The other investigator, who did not know how long the child inhaled in the morning, evaluated pain and vital signs 1 and 30 minutes after the child returned to bed.

DETAILED DESCRIPTION:
This randomized clinical trial research experimental design was performed with pediatric burn patients on May 2018-May 2019. Routine treatment of any child was not interfered with during the data collection phase of the study.

Sample

The minimum sample size in each intervention and control group was considered 36 using G power formula with a = 0.05, power of 80%, 95% confidence interval (Gpower 3.1.9.2., Germany). Allocation to the groups was performed using the Stratified Randomization. The absence of differences in age, vital signs and pain levels between groups prior to the intervention was achieved using Stratified Randomization method.

Intervention Protocols

In the clinic where the study was conducted, all children are routinely given hydrotherapy treatment for the examination of the burn area as of 10 am every morning and then dressings are applied.

Besides routine care, the Control Group was treated with jojoba oil (Simmondsia Chinensis- produced by Arifoğlu, obtained from jojoba fruits by cold squeezing method) inhalation aromatherapy 15 minutes before Hydrotherapy. Jojoba oil was used as a placebo because it had no specific odour. Besides routine care, Intervention-15 Group received lavender oil (Lavandula angustifolia Miller Oleum-produced by Arifoğlu, obtained from lavender flowers by water vapour distillation method) inhalation aromatherapy 15 minutes before Hydrotherapy and besides routine care, Intervention-60 Group received lavender oil inhalation aromatherapy 60 minutes before Hydrotherapy. 0.5 ml (8.44 minim-imperial) of aromatherapy oil, which had been dripped into 7.5x7.5 cm gauze 15 or 60 minutes before the start of Hydrotherapy, was placed 20 cm (7.87 inches) away from the child's nose by the clinical nurse. To conceal the allocation, the group in which the child belongs is only known to the clinical nurse who has placed the aromatherapy oil-soaked gauze in the child's room and this clinical nurse did not carry out any assessment of the child's outcomes.

Data Collection

Before randomization, the characteristics of all participants were collected using the Turkish version of the FLACC Pain Scale, Demographic Data Collection Form, and the Vital Signs Follow-up Form which were developed by the researchers.

By the clinical nurse 0.5 ccs of aromatherapy oil, which had dripped into the gauze, was placed 20 cm away from the child's nose. The child who inhaled the oil was then taken to hydrotherapy and then dressing. The pain and vital signs of the child were evaluated and recorded 1 minute and 30 minutes after the child returned to bed by a researcher who was blind to the study groups.

ELIGIBILITY:
Inclusion Criteria:

* aged 2 months-7 years,
* having a second degree of superficial burn,
* willing to participate in the study,
* receiving hydrotherapy application (wet dressing),
* dressing the child with the same dressing material,
* having no chronic pain,
* having scalding burn,
* having no surgery record to treat burns,
* having no pathogen reproduction at the burn area,
* having no stage of epitheliazation,
* having analgesic therapy containing the same active substance.

Exclusion Criteria:

-

Ages: 2 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
mean arterial pressure | 1 day
  The mean arterial pressure of the child was evaluated and recorded before dressing, also 1 and 30 minutes after the dressing.
body temperature | 1 day
  The body temperature of the child was evaluated and recorded before dressing, also 1 minute and 30 minutes after the dressing.
heart rate | 1 day
  The heart rate of the child was evaluated and recorded before dressing, also 1 minute and 30 minutes after the dressing.
respiratory rate | 1 day
  The respiratory rate of the child was evaluated and recorded before dressing, also 1 minute and 30 minutes after the dressing.
FLACC Pain Scale Scores | 1 day
  The FLACC Pain Scale scores of the child was evaluated and recorded before dressing, also 1 minute and 30 minutes after the dressing.
  FLACC (The Face, Legs, Activity, Cry, Consolability Scale) Pain Scale used by Merkel et al in 1997 in children between 2 months-7 years of age. With this scale, five behavioral criteria such as facial expression, the position of legs, movements, crying and comforting are evaluated. Each episode is rated 0-2 with scores ranging from 0-10 in total, the lower the score, the less pain is said .0 points:" no pain "1-3 points:" there is little pain "4-6 points:" there is moderate pain " 7-10 points:" there is much pain".

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Behcet Uz Children's Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No